CLINICAL TRIAL: NCT00767741
Title: Evaluation of the Effects of Heating or Massaging or Vibrating at the Vicinity of the Insulin Delivery Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: INS-0417-08-HMO
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes
Keywords: diabetes; post prandial glucose level; insulin; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- with treatment (Experimental)
  Interventions: Device: with heat and massage

INTERVENTIONS:
Device: with heat and massage — For the with intervention group a treatment to the injection site is applied after each insulin bolus injection.

SUMMARY:
The aim of this study is to test the pharmacodynamics of insulin analogs and their dependence on external and physiological alterations. We plan to compare the pharmacodynamics of insulin analog delivery in regular conditions and in the presence of increased perfusion of the delivery site, achieved by way of local warming and movement

ELIGIBILITY:
Inclusion Criteria:

1. Participant age between 18- 65 years old
2. Type I or Type II diabetes
3. HbA1c 6-12%
4. Does not suffer from sever hypertension, kidney, liver or heart disease
5. Does not suffer from active Ischemic heart disease
6. Is willing to sign the consent form

Exclusion Criteria:

1. Participants age < 18 or > 65
2. Pregnancy
3. Breast feeding women
4. Un-controlled diabetes, HbA1c values > 12% range
5. Suffers from active Ischemic heart disease
6. Alcohol addiction
7. Is not prepared to signed the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Insulin blood level with and with out the intervention | at the end of every daily study

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical center, Jerusalem, Other, Israel